CLINICAL TRIAL: NCT02997423
Title: Prospective Phase II Study of Cytochrome C Oxidase Activity as a Novel Biomarker In Subjects With Newly Diagnosed Primary Glioblastoma Multiforme
Brief Title: Cytochrome C Oxidase Activity in Newly Diagnosed Glioblastoma Multiforme (GBM)
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); NeuroNEXT Network (Other)
Responsible Party: Principal Investigator, Corinne Griguer, Associate Professor, University of Iowa
Other Study IDs: NN106; U01NS093663 (NIH)
Record Dates: First submitted 2016-12-09; First posted 2016-12-20 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Glioblastoma
Keywords: Glioblastoma Multiforme; Biomarker; Cytochrome C Oxidase; Newly diagnosed
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue and DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-institutional, consortium-based, non-interventional prospective blinded endpoints clinical study to determine whether high activity of Cytochrome C Oxidase (CcO) in tumor specimens from subjects with newly diagnosed primary GBM is associated with shortened OS (primary outcome) and PFS (secondary outcome) times.

DETAILED DESCRIPTION:
This Biomarker trial is designed to prospectively evaluate the hypothesis that the overall survival (OS) time of a subject with newly diagnosed primary GBM tumors, treated by standard of care (SOC), is a function of the CcO enzymatic activity in the tumor (OS; time interval from date of first diagnosis to death from any cause, irrespective of post-SOC therapies, assessed up to 24 months from accrual). In particular, tumors with high CcO activity are associated with shorter OS time as compared to tumors with low CcO activity. SOC consists of post-surgical radiation therapy with concurrent Temozolomide followed by up to 12 cycles of adjuvant Temozolomide.

Additional outcomes are to study the relation between CcO activity in the GBM tumors and progression free survival times (PFS; time intervals from dates of diagnosis to documented disease progression by MRI or tumor-related death) and, to compare the prognostic abilities of CcO activity to other frequently used biomarkers, namely the methylation status of O6-methylguanine-DNA methyltransferase (MGMT), on OS and PFS.

Tumor tissue will be submitted by participating centers for measurements of the CcO/Citrate Synthase (CS), MGMT promoter methylation. The subjects will agree to receive the SOC treatment. The therapeutic option at the time of first recurrence is at the discretion of the treating physician. PFS and OS times will be compared with high vs. low CcO activity and with the MGMT methylation status of the tumor. At the time of death or at 24 months s/p enrollment (whichever comes first), the site PI will complete an exit form documenting the details of enrollees' treatment history and date(s) of any tumor progression.

ELIGIBILITY:
Inclusion Criteria

1. Willingness and ability to provide written informed consent and to comply with the study protocol as judged by Physician interview (NOTE: This could be patient's Neurosurgeon, Neuro-Oncologist or Study Investigator). If patient lacks capacity to consent, a legally authorized representative is allowed to provide written informed consent.
2. Age ≥ 21 years
3. Karnofsky Performance Status (KPS) ≥ 60.
4. Subjects' planned upfront treatment to be standard of care treatment with radiotherapy and temozolomide (i.e. TEMODAR) for histologically confirmed GBM at initial diagnosis
5. No history of other malignancies except adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, or other curatively treated solid tumors with no evidence of disease for at least 5 years.
6. No serious active infection (e.g., wound infection requiring parenteral antibiotics) or other serious underlying medical conditions that in the opinion of the investigator would compromise standard of care treatment.
7. No other condition (e.g., psychological or geographical) that would preclude study compliance.
8. An MRI that is consistent with a primary malignant glioma
9. Histologically confirmed newly diagnosed primary GBM before treatment using World Health Organization (WHO) classification criteria (A local pathology report constitutes adequate documentation of histology for initial study enrollment, however central pathology review will be required to confirm the diagnosis of GBM for final data analysis).
10. Viability of tumor tissue representative of GBM ≥ 70 mg, snap-frozen within 30 minutes of resection, 10 minutes or less at room temperature.
11. All subjects must have received maximal safe resection followed by standard radiation therapy with concomitant Temozolomide taken during the course of radiation therapy.

Exclusion Criteria:

Exclusion criteria are proposed that will exclude subjects with pre-existing co-morbidities that could contribute to pre-mature death (e.g., significant cardiovascular history), with non-included pretreated tumors occupying either intracranial and extra-axial space, significantly impaired neurological performance status (e.g., KPS>60), with glial tumors that are genomically distinct from primary GBM tumors (e.g., gliomas arising from a previously diagnosed lower grade than GBM) or those unable to complete the fundamental requirements of the study.

1. Inability to fulfill the requirements of the protocol
2. Secondary GBM or other gliomas.
3. History of sensitivity to Temozolomide.
4. Planned upfront treatment with any anti-angiogenic agent targeting the (vascular endothelial growth factor (VEGF) pathway including but not limited to bevacizumab, cediranib, vandetanib, sunitinib, pazopanib, aflibercept, or sorafenib or any immunotherapy regimen.
5. Any severe post-operative infection or other complications that may significantly delay the initiation of brain tumor therapy, or other conditions that, in the opinion of the investigator, would compromise the subject's ability to participate in the study.

Note: Use of Gliadel wafers, in combination with surgical resection, is allowed if the patient is to follow standard-of-care treatment post-operatively (i.e., radiation therapy with temozolomide). Use of Gliadel wafers during surgery with only radiation therapy post-operatively is excluded (i.e., omitting temozolomide).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed primary Glioblastoma multiforme (GBM) patients who will receive standard of care treatment.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Date of diagnosis through 24 months after enrollment
  This biomarker trial is designed to prospectively evaluate the hypothesis that the overall survival (OS) time of a subject with newly diagnosed primary GBM tumors, treated by standard of care (SOC), is a function of the CcO enzymatic activity in the tumor. OS is defined as the time interval from date of first diagnosis to death from any cause, irrespective of post-SOC therapies, assessed up to 24 months from accrual.

OTHER OUTCOMES:
Progression Free Survival (PFS) | Date of diagnosis through 48 months after enrollment
  This biomarker trial is designed to prospectively evaluate the hypothesis that progression free survival time (PFS) is a function of the CcO enzymatic activity in the tumor. PFS is defined as time interval from date of surgery to first documented progression according to the RANO criteria, irrespective of post-SOC therapies.
MGMT methylation status on OS and PFS | Date of diagnosis through 24 months after enrollment
  Compare the prognostic abilities of CcO activity to another frequently used biomarker, the methylation status of O6-methylguanine-DNA methyltransferase (MGMT) on OS and PFS times.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne E Griguer, PhD, Principal Investigator — University of Iowa
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UC Davis, Sacramento, California
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University Medical School, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Stony Brook, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Swedish Neuroscience Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The requestor must submit a formal written request for data sharing, and the request must be approved by the NeuroNEXT Steering Committee and the Publication Committee before any data are shared. Prior to data sharing, the DCC and the external source must also execute a data sharing agreement that includes a description of the data that are requested and how the data will be shared. A contract / usage agreement may be required.
  The DCC will submit de-identified datasets and associated documentation to NINDS for archiving and public access, consistent with the current NINDS Data Sharing policy. The DCC will provide documentation with each final dataset to ensure that other users can efficiently and accurately use the dataset, and to prevent misinterpretation or misuse. This documentation may include information about how the data were collected, provide details about the code used to generate the dataset, and define variables and variable field locations.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Upon request.
Access Criteria: Written request to principal investigator.

REFERENCES:
- [Background] Vogelbaum MA, Jost S, Aghi MK, Heimberger AB, Sampson JH, Wen PY, Macdonald DR, Van den Bent MJ, Chang SM. Application of novel response/progression measures for surgically delivered therapies for gliomas: Response Assessment in Neuro-Oncology (RANO) Working Group. Neurosurgery. 2012 Jan;70(1):234-43; discussion 243-4. doi: 10.1227/NEU.0b013e318223f5a7. PMID 21593697
- [Background] Galanis E, Wu W, Cloughesy T, Lamborn K, Mann B, Wen PY, Reardon DA, Wick W, Macdonald D, Armstrong TS, Weller M, Vogelbaum M, Colman H, Sargent DJ, van den Bent MJ, Gilbert M, Chang S. Phase 2 trial design in neuro-oncology revisited: a report from the RANO group. Lancet Oncol. 2012 May;13(5):e196-204. doi: 10.1016/S1470-2045(11)70406-5. PMID 22554547
- [Result] Griguer CE, Oliva CR, Coffey CS, Cudkowicz ME, Conwit RA, Gudjonsdottir AL, Ecklund DJ, Fedler JK, Neill-Hudson TM, Nabors LB, Benge M, Hackney JR, Chase M, Leonard TP, Patel T, Colman H, de la Fuente M, Chaudhary R, Marder K, Kreisl T, Mohile N, Chheda MG, McNeill K, Kumthekar P, Dogan A, Drappatz J, Puduvalli V, Kowalska A, Graber J, Gerstner E, Clark S, Salacz M, Markert J. Prospective biomarker study in newly diagnosed glioblastoma: Cyto-C clinical trial. Neurooncol Adv. 2021 Dec 24;4(1):vdab186. doi: 10.1093/noajnl/vdab186. eCollection 2022 Jan-Dec. PMID 35088051